CLINICAL TRIAL: NCT00465426
Title: Assessment of Cardiovascular Risk in HIV Patients
Brief Title: HIV and Cardiovascular Risk
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Steven K. Grinspoon, MD, Principal Investigator, Massachusetts General Hospital
Other Study IDs: DK49302-10AR; R01DK049302 (NIH)
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: HIV Infections; Cardiovascular Disease
Keywords: HIV Infection; Cardiovascular Disease; Antiretroviral Therapy; Inflammatory Markers; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood will be frozen for end of study analysis for insulin, CRP, adiponectin, TNF-α, sTNFR2, IL-6, PAI-1, MCP-1
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: HIV Positive men and women 18-65 years of age
- 2: HIV negative men and women 18-65 years of age

SUMMARY:
HIV-infected patients treated with combination antiretroviral therapy demonstrate metabolic abnormalities that may predispose them to cardiovascular disease. In HIV-infected patients we will investigate progression rates of cardiovascular disease and assess whether these progression rates are predicted by increased inflammatory indices.

DETAILED DESCRIPTION:
HIV-infected patients treated with combination antiretroviral (ARV) therapy increasingly demonstrate metabolic abnormalities, including dyslipidemia, insulin resistance and body composition abnormalities that may predispose them to cardiovascular disease (CVD). Initial studies suggest increased carotid intima-media thickness (IMT) and endothelial dysfunction in this population. Increased carotid IMT over time has been demonstrated in HIV-infected patients compared to control subjects. However, traditional risk factors, such as dyslipidemia, diabetes mellitus and body composition changes alone do not fully predict increased cardiovascular disease in HIV-infected patients. One possible explanation is increased inflammation, related directly to effects of ARV therapy or indirectly from changes in fat distribution. In preliminary studies, our group has shown that changes in fat distribution were highly predictive of TNF and IL-6, as well as adiponectin, and that specific inflammatory cytokines were related in cross-sectional studies to increased IMT. In the proposed study we will investigate using detailed methodologies the relationship between adipocytokine concentrations and subclinical atherosclerosis in both cross-sectional and longitudinal studies. We will determine in HIV-infected patients on ARVs for greater than 6 months, progression rates of IMT and whether progression rates are predicted by increased inflammatory indices, controlling for traditional risk factors, and body composition changes. We will test the hypothesis that inflammation, more than traditional risk factors and ARV use, mediates subclinical atherosclerotic disease in HIV-infected patients.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Group 1 (HIV-infected group)

1. Age greater than or equal to 18 and less than or equal to 65 years of age
2. HIV positive, on the same combination ARV regimen for > than 6 months, including but not limited to either 2 NRTIs and an NNRTI or PI, or a triple NRTI regimen
3. CD4 >350 cells/mm3

Inclusion Criteria for Group 2 (HIV Negative, Healthy Control, age and BMI matched to HIV subjects)

1. No history of HIV infection (negative HIV test)
2. Age greater than or equal to 18 and less than or equal to 65 years of age

Exclusion Criteria:

Exclusion Criteria for Group 1 (HIV-infected group)

1. Hgb < 10.0 g/dL, creatinine > 1.5 mg/dL, SGPT > 2.5x ULN
2. Use of glucocorticoid, testosterone, growth hormone or other anabolic agents within the past 6 months
3. New antiretroviral regimen within 6 months of study initiation
4. Active substance abuse
5. Medications known to affect glucose or body composition
6. Positive pregnancy test or recently pregnant within the past year or lactating
7. Presence of active cancers
8. Acute viral, bacterial or other infections (excluding HIV)
9. Weight loss in the past 3 months of greater than 10 pounds

Criteria for Group 2 (HIV Negative, Healthy Control, age and BMI matched to HIV subjects)

1. Hgb < 10.0 g/dL, creatinine > 1.5 mg/dL, SGPT > 2.5x ULN
2. Use of glucocorticoid, testosterone, growth hormone or other anabolic agents within the past 6 months.
3. Active substance abuse
4. Medications known to affect glucose or body composition
5. Positive pregnancy test or recently pregnant within the past year or lactating
6. Acute viral, bacterial or other infections
7. Weight loss in the past 3 months of greater than 10 pounds

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Flyers and advertisements regarding this study will be posted in community centers and newspapers
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2007-04; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Carotid Intima Media Thickness | 2 years
Waist Circumference | 2 years
Blood pressure | 2 years
Lipid levels | 2 years
Glucose | 2 years

SECONDARY OUTCOMES:
Inflammatory markers | 2 years
Visceral adiposity | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven K Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Fitch KV, Stavrou E, Looby SE, Hemphill L, Jaff MR, Grinspoon SK. Associations of cardiovascular risk factors with two surrogate markers of subclinical atherosclerosis: endothelial function and carotid intima media thickness. Atherosclerosis. 2011 Aug;217(2):437-40. doi: 10.1016/j.atherosclerosis.2011.04.009. Epub 2011 Apr 16. PMID 21570076